CLINICAL TRIAL: NCT05003258
Title: Functional and Anatomical Outcomes of Dexamethasone Intra-vitreal Implant in Patients with Resistant Macular Edema Secondary to Retinal Vein Occlusion After Intravitreal Anti-VEGF Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menatallah Gamal Saleh, Assistant lecturer of Ophthalmology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAODIIPMERVO
Record Dates: First submitted 2021-07-15; First posted 2021-08-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2023-10

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: Dexamethasone Intravitreal Implant; Retinal vein occlusion; Macular Edema
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with RVO (Other): Dexamethasone Intravitreal Implant is used in patients with Macular ar edema due to retinal vein occlusion either from the start or after unsatisfactory response to anti - VEGF
  Interventions: Device: Intravitreal injection of Dexamethasone implant

INTERVENTIONS:
Device: Intravitreal injection of Dexamethasone implant — Intravitreal injection of Dexamethasone implant
  Other Names: Ozurdex

SUMMARY:
Retinal vein occlusion (RVO) is one of the most common causes of vision loss due to retinal vascular disease. Incidence of RVO has been raised in the last years due to increased coexisting systemic vascular risk factors as arterial hypertension, obesity, diabetes mellitus and COVID-19. Macular edema (ME) is a major sight-threatening complication of branch retinal vein occlusion (BRVO) and central retinal vein occlusion (CRVO). BRVO and CRVO have the same pathology, an elevation in the intravascular pressure in the occluded vein leading to vascular wall damage causing leakage of fluid and release of inflammatory cytokines as vascular endothelial growth factor (VEGF), respectively.

In the past, the standard treatment for BRVO-related ME was grid laser photocoagulation and for CRVO-related ME was observation. But subsequent randomized controlled trials demonstrated significant functional and anatomical improvements among patients with ME secondary to BRVO or CRVO treated with intravitreal injections of vascular endothelial growth factor (VEGF) inhibitors or corticosteroids compared to those treated with laser only. Anti-VEGF therapy decrease intravenous pressure, enhance blood flow and improve venous diameter and tortuosity. Also, intravitreal corticosteroid injection has been shown to improve vision and central macular thickness (CMT).

Dexamethasone intravitreal implant (Ozurdex®, Allergan Inc., Irvine, CA, USA) has potent antiangiogenic and anti-inflammatory effects. Also it decreases the vascular permeability playing an important role in treating ME secondary to RVO. However, majority of eyes have been treated previously then shifted to dexamethasone implant as a second line for treatment of refractory RVO related ME.

DETAILED DESCRIPTION:
Aim of the research is To evaluate functional and anatomical outcomes of ozurdex injection in patients with RVO related macular edema.

And evaluation of the safety of ozurdex injections regarding intraocular pressure increase, cataract development or endophthalmitis.

Type of the study: Interventional Case Series. Study Setting: Assiut University Hospital (Ophthalmology Department).

Study subjects:

1. Inclusion criteria:

   1. Patients with macular edema secondary to BRVO and CRVO.
   2. Presence of macular edema >3oo μ on OCT evaluation.
   3. visual acuity of +0.3 logarithm of the minimum angle of resolution (logMAR) or worse.
2. Exclusion criteria:

   1. Presence of coexisting retinal disease (such as diabetic retinopathy, age related macular degeneration, vitreo-macular traction, or epiretinal membrane).
   2. Media opacities (cataract) that could decrease visual acuity (VA).
   3. Previous ocular trauma or vitreoretinal surgery.
   4. Patients with glaucoma or known to be steroid responders.

Baseline evaluation:

1. Complete ophthalmic evaluation including assessment of distance BCVA using Snellen charts and will be converted to logarithm of the minimum angle of resolution (logMAR), tonometry, slit-lamp bio microscopy, gonioscopy and dilated fundus examination.
2. Thorough clinical history and review of other systems involvement as well as full drug history.

Imaging:

SD-OCT (Spectralis; Heidelberg Engineering, Heidelberg, Germany) with automated CMT measurements through a dilated pupil.

Color fundus photography and fluorescein angiography will be performed for every patient at baseline to document the clinical appearance and type of RVO using Topcon TRC-NW8F (Topcon Medical Systems, Inc., Tokyo, Japan).

OCTA will be performed before and after injection.

Outcome measures:

Primary (main):

* Assessment of VA and CMT improvement after use of dexamethasone implant in macular edema secondary to RVO.
* Evaluation the safety of intravitreal Ozurdex injection regarding adverse events as IOP increase, cataract development or endophthalmitis.

  b. Secondary (subsidiary):
* To evaluate the incidence and onset of occurrence of any adverse event or recurrence.
* To correlate between BCVA and CMT throughout the duration of the study. Data collection: data will recorded in the form of excel spreadsheets. Computer software: SPSS. Statistical tests: Tests of normality will be performed, if data are normally distributed student t-test will be done and if not, Mann-Whitney test will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients with macular edema secondary to BRVO and CRVO.
* Presence of macular edema >3oo μ on OCT evaluation.
* visual acuity of +0.3 logarithm of the minimum angle of resolution (logMAR) or worse.

Exclusion Criteria:

* Presence of coexisting retinal disease (such as diabetic retinopathy, age related macular degeneration, vitreo-macular traction, or epiretinal membrane).
* Media opacities (cataract) that could decrease visual acuity (VA).
* Previous ocular trauma or vitreoretinal surgery.
* Patients with glaucoma or known to be steroid responders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
_Assessment of VA using snellen chart after use of ozurdex in macular edema secondary to RVO. | 2 years

SECONDARY OUTCOMES:
- To evaluate the incidence and onset of occurrence of any adverse event or recurrence. | 2 years
  Safety of intravitreal Ozurdex injection

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Asyut, Egypt

REFERENCES:
- [Background] Teja S, Sawatzky L, Wiens T, Maberley D, Ma P. Ozurdex for refractory macular edema secondary to diabetes, vein occlusion, uveitis and pseudophakia. Can J Ophthalmol. 2019 Oct;54(5):540-547. doi: 10.1016/j.jcjo.2018.12.005. Epub 2019 Jan 25. PMID 31564342
- [Background] Maggio E, Mete M, Maraone G, Attanasio M, Guerriero M, Pertile G. Intravitreal Injections for Macular Edema Secondary to Retinal Vein Occlusion: Long-Term Functional and Anatomic Outcomes. J Ophthalmol. 2020 Feb 13;2020:7817542. doi: 10.1155/2020/7817542. eCollection 2020. PMID 32104597